CLINICAL TRIAL: NCT00000664
Title: Safety and Efficacy of Polyethylene Glycolated IL-2 (PEG IL-2) Plus Zidovudine in HIV Positive, Asymptomatic and Symptomatic Individuals
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Model: Parallel | Purpose: Treatment
Other Study IDs: ACTG 141; CS-PG89-36; FDA 70A
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2008-08-04 (Estimated); Status verified 1994-12

CONDITIONS: HIV Infections
Keywords: Polyethylene Glycols; Interleukin-2; Drug Evaluation; Zidovudine
MeSH Terms: conditions — HIV Infections | interventions — Interleukin-2; Zidovudine

INTERVENTIONS:
Drug: Interleukin-2, Polyethylene Glycolated
Drug: Zidovudine

SUMMARY:
To determine the safety of polyethylene glycolated IL-2 (PEG IL2) administered weekly or biweekly (per amendment) in a setting of oral zidovudine (AZT). To determine the effect of PEG IL2 in combination with AZT on parameters assessing the immune system as well as HIV virus and antibody titers. To evaluate a chronic dosing study phase offered to patients who complete the initial 25-week regimen.

Recent research has focused on enhancing cell-mediated immunity and reducing or eliminating viral replication (reproduction and growth). A main thrust of current treatment is the combination of antiviral drugs that may be more effective when combined than when each is used alone.

DETAILED DESCRIPTION:
Recent research has focused on enhancing cell-mediated immunity and reducing or eliminating viral replication (reproduction and growth). A main thrust of current treatment is the combination of antiviral drugs that may be more effective when combined than when each is used alone.

Four groups are studied for a period of at least 25 weeks. Patients are observed for a minimum of 6 hours after infusion of PEG IL2. The 4 groups of patients are: Group A - asymptomatic with T4 count > 400 cells/mm3 (7 patients); Group B - asymptomatic with T4 count between 200 and 400 cells/mm3 (7 patients); Group C - asymptomatic with T4 count < 200 cells/mm3 (5 patients); Group D - diagnosed as having AIDS related complex (ARC) or AIDS (7 patients). All patients receive AZT. After a minimum 2-week period of AZT, patients receive an infusion of PEG IL-2 at 3 consecutive weekly intervals, followed by a 3-week period of AZT alone. This cycle (3 weeks of AZT and PEG IL-2 followed by 3 weeks of AZT alone) is repeated a total of three times (for a total of 18 weeks) followed by 8 weeks of AZT alone.

PER AMENDMENT: Ten patients may qualify for one of two groups: Group 1 - T4 count 200 - 400 cells/mm3 and meet all criteria established for Group B of the original protocol; Group 2 - T4 count < 200 cells/mm3 and meet all criteria established for Groups C and D of original protocol. Patients will receive an amended schedule of PEG IL2 IV every other week for eight doses, with dose escalation every other week for eight weeks permitted only in Group 2 patients who failed to show a 20 percent rise in T4 count at week 9 and who suffered no CNS or other adverse events at the lower dose.

PER ADDITIONAL AMENDMENT: Up to 10 additional patients may be treated at each dose of PEG IL2 on the biweekly schedule. Patients who respond to treatment on the biweekly schedule are eligible for an additional 9 weeks at their current dose.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Prophylactic pentamidine for Pneumocystis carinii pneumonia (PCP).
* Topical steroids.

Patients must:

* Be HIV positive. Fit one of the zidovudine use groups listed in Disease Status. Be able to give informed consent.

Allowed:

* Basal cell carcinoma of the skin, in situ carcinoma of the cervix, Kaposi's sarcoma.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Major organ allograft.
* Significant cardiac disease or central nervous system lesions.
* Known previous intolerance to zidovudine (AZT) at 500 mg/day.
* Active opportunistic infections. Score of > 0.5 on the ACTG AIDS dementia complex staging test. Any focal abnormality on neurologic exam.

Concurrent Medication:

Excluded:

* Chemotherapy, hormonal therapy, or other immunotherapy.
* Other investigational drugs, agents, or devices.
* Beta-blockers.
* Steroids other than topical.
* Antihypertensive medication other than diuretics.

Concurrent Treatment:

Excluded:

* Radiation therapy.

Patients with the following are excluded:

* History of seizures. Concurrent neoplasms not specifically allowed.
* Concomitant conditions listed in Exclusion Co-existing Conditions.

Prior Medication:

Excluded within 30 days prior to study entry:

* Anti-HIV medication other than zidovudine (AZT).
* Immunomodulators.
* Systemic steroids.
* Interferons.
* Interleukins.
* Other chemotherapy.

Prior Treatment:

Excluded within 30 days prior to study entry:

* Radiation therapy.

Excluded within 4 weeks prior to study entry:

* Groups B, C, D
* Transfusions.

Active substance abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26

CONTACTS AND LOCATIONS:
Overall Officials: TC Merigan, Study Chair; J Korvick, Study Chair
Locations (1):
- Stanford Univ School of Medicine, Stanford, California, United States

REFERENCES:
- [Background] Wood R, Montoya JG, Kundu SK, Schwartz DH, Merigan TC. Safety and efficacy of polyethylene glycol-modified interleukin-2 and zidovudine in human immunodeficiency virus type 1 infection: a phase I/II study. J Infect Dis. 1993 Mar;167(3):519-25. doi: 10.1093/infdis/167.3.519. PMID 8095058